CLINICAL TRIAL: NCT00739622
Title: A Phase I, Open-label Drug-drug Interaction Trial to Investigate the Effect of TMC278 25 mg q.d. on the Steady State Pharmacokinetics of Ethinylestradiol and Norethindrone, in Healthy Women
Brief Title: TMC278-TiDP6-C136: Effect of TMC278 on Ethinylestradiol and Norethindrone in Healthy Women.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tibotec Pharmaceuticals, Ireland (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR010762
Record Dates: First submitted 2008-08-20; First posted 2008-08-22 (Estimated); Last update posted 2010-04-28 (Estimated); Status verified 2010-04

CONDITIONS: HIV; AIDS; Oral Contraceptive
Keywords: TMC278-TiDP6-C136; TMC278-C136; Healthy Volunteer
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Rilpivirine

INTERVENTIONS:
Drug: TMC278

SUMMARY:
The purpose of this study is to investigate the pharmacokinetic interaction between the combination of ethinylestradiol and norethindrone and TMC278 25 mg once daily. Pharmacokinetics means how the drug is absorbed into the bloodstream, distributed in the body and eliminated from the body. Furthermore the short-term safety and tolerability (how well the body tolerates the drug) of co-administration of TMC278 and ethinylestradiol and norethindrone, in healthy women, will be assessed.

DETAILED DESCRIPTION:
Human immunodeficiency virus (HIV)-infected patients are routinely being treated with combinations of 3 or 4 drugs (highly active antiretroviral therapy [HAART]), to reduce the risk of viral resistance development. Development of new potent antiretroviral (ARV) drugs is urgently needed to prolong suppression of viral replication in patients infected with HIV. This is a Phase I, open-label trial in healthy women to investigate the pharmacokinetic interaction between the combination of ethinylestradiol and norethindrone and TMC278 25 mg once daily. The trial aims to allow further recommendations regarding the concurrent use of oral contraceptives and TMC278. The trial population will consist of 18 healthy women who are stable on oral contraceptives (OC), specifically ethinylestradiol and norethindrone, or who, if they are not currently using this OC, are willing to start or switch to this OC for the duration of the study.

Healthy volunteers will receive the OC once daily for 21 days for at least 1 OC cycle prior to Day 1 [stabilizing OC cycle from Day -28 to Day -1]. During the second OC cycle [from Day 1 to Day 28], subjects will receive the OC alone once daily for 21 days [Treatment A]. During the third OC cycle [from Day 29 to 56], subjects will receive the OC once daily for 21 days and in addition TMC278 25 mg q.d. in the morning for 15 days, starting on the first day of OC intake (Day 29) [Treatment B]. Full 24-hour pharmacokinetic profiles of ethinylestradiol and norethindrone will be determined after the first 2 weeks of the second OC cycle (Treatment A: OC alone; Day 15) and after the first 2 weeks of the third OC cycle (Treatment B: OC+TMC278; Day 43). A full 24-hour pharmacokinetic profile of TMC278 will be determined on Day 43. Blood samples on these days will be drawn just before drug intake (predose), and at 0.5, 1, 1.5, 2, 3, 4, 5 (Day 43 only), 6, 9, 12, 16 (Day 43 only) and 24 hours postdose. Safety evaluations include evaluation of adverse events, physical examination including vital signs, ECGs and laboratory hematology and biochemistry assessments. Healthy volunteers will receive a tablet of ethinylestradiol and norethindrone OC once daily for 21 days for at least 1 OC cycle prior to Day 1. During the second OC cycle, healthy volunteers will receive a tablet of ethinylestradiol and norethindrone OC alone once daily for 21 days. During the third OC cycle, healthy volunteers will receive a tablet of ethinylestradiol and norethindrone once daily for 21 days and in addition a tablet of TMC278 25 mg once daily in the morning for 15 days.

ELIGIBILITY:
Inclusion Criteria:

* Willing to start or continue oral contraceptive therapy, specifically ethinylestradiol and norethindrone, for the duration of the study
* Consent to a method of birth control in addition to the OC trial medication
* Non-smoking or smoking no more than 10 cigarettes, or 2 cigars, or 2 pipes per day for at least 3 months prior to screening
* Body Mass Index (BMI) of 18.0 to 30.0 kg/m2, extremes included
* Healthy on the basis of a physical examination, medical history, electrocardiogram, vital signs and the results of blood biochemistry and hematology tests and a urinalysis carried out at screening.

Exclusion Criteria:

* The most important eligibility criteria are: Not pregnant or breastfeeding
* Not postmenopausal
* No positive HIV test
* No alcohol or barbiturate, amphetamine, recreational or narcotic drug use
* No hepatitis A, B or C infection
* No currently active gastrointestinal, cardiovascular, neurologic, psychiatric, metabolic, renal, hepatic, respiratory, inflammatory or infectious disease
* No history of significant skin disease
* No previously demonstrated clinically significant allergy or hypersensitivity to any of the excipients of the medication administered in this trial (i.e. TMC278, Ovysmen®)
* No clinical significant abnormal finding in the gynaecological examination
* No currently active gynaecological disorders
* No major medical condition that would preclude the safe administration of oral contraceptive therapy
* No participation in an investigational drug trial within 60 days prior to the start of the first OC cycle

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2008-07; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study is to determine the effect of steady-state concentrations of TMC278 25 mg once daily on the steady-state pharmacokinetics of ethinylestradiol 35 mcg and norethindrone 1 mg once daily.

SECONDARY OUTCOMES:
The secondary objective of this study is to evaluate the short-term safety and tolerability of coadministration of TMC278 and ethinylestradiol and norethindrone OC in healthy women.

CONTACTS AND LOCATIONS:
Overall Officials: Tibotec Pharmaceuticals Limited Clinical Trial, Study Director — Tibotec Pharmaceutical Limited

REFERENCES:
- [Derived] Crauwels HM, van Heeswijk RP, Buelens A, Stevens M, Hoetelmans RM. Lack of an effect of rilpivirine on the pharmacokinetics of ethinylestradiol and norethindrone in healthy volunteers. Int J Clin Pharmacol Ther. 2014 Feb;52(2):118-28. doi: 10.5414/CP201943. PMID 24161160